CLINICAL TRIAL: NCT06307028
Title: Sistas Informing Sistas on Topics About AIDS and Prevention
Brief Title: Sistas Informing Sistas on Topics About AIDS and Prevention (SISTA-P)
Acronym: SISTA-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Shawnika J. Hull, PhD, Associate Professor, Department of Communication, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro2023002116; K01DA050496 (NIH)
Record Dates: First submitted 2024-02-23; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Health Behavior, Risky; Health Knowledge, Attitudes, Practice; Health-Related Behavior
Keywords: Black women; HIV
MeSH Terms: conditions — Health Risk Behaviors; Behavior; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SISTA-P Intervention (Experimental): Participants will complete four sessions lasting up to three hours each over the course of one week. The sessions will be overseen by two facilitators and a technical monitor. Core elements of SISTA-P are: (1) small group discussions, modeling and role-play that facilitate repetition, reinforcement and sequential approximation; (2) skilled facilitators; (3) gender and culturally specific materials to enhance pride and self-worth; (4) teaching negotiation, self-advocacy; and (5) HIV prevention relevant skills; (6) discussing gender and culture-specific barriers and facilitators to prevention; and (7) enhancing HIV prevention norms and self-efficacy. Each discussion group will consist of 12- 15 participants and each cycle will consist of one group. Participants will be asked to complete a follow up survey and two booster sessions. They will also be asked to submit photo-confirmation of PrEP prescription to the research team.
  Interventions: Behavioral: SISTA-P Intervention

INTERVENTIONS:
Behavioral: SISTA-P Intervention — This intervention is a small group discussion designed specifically for Black women. The sessions cover topics including: self pride and self-care; HIV & PrEP education; assertiveness skills training; coping skills; skills practice; and barriers and facilitators to HIV prevention and PrEP.

SUMMARY:
In this project, the investigators will provide a new HIV prevention training and empowerment sessions to Black women in Washington D.C. who are at high risk for getting HIV. This training is tailored to the experience of Black women and seeks to reduce the high HIV transmission rates in the Black community.

DETAILED DESCRIPTION:
Experienced facilitators will implement two cycles of six 3-hour sessions with up to 15 participants per cycle while expert panelists observe. After each session, participants and subject matter expert observers will complete brief surveys. Surveys following each session include closed and open-ended measures: six items rating how well the session conveyed core information (e.g., I am confident I can communicate more effectively [Session 3]; I have a better understanding of the effects of alcohol on making sexual choices, [Session 4]) and single-item scales to evaluate the facilitator's performance and the session overall. In open-ended measures, respondents will be prompted to elaborate on their survey responses to identify ways the session could be improved.

ELIGIBILITY:
Inclusion Criteria:

* Black women are eligible if you:
* Have sex with men
* Are age 18+
* Live in Washington D.C.
* Are not HIV+

Exclusion Criteria:

* HIV+

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Black women are eligible for this study.
Enrollment: 30 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention Scale | At the end of each cycle (each cycle is 42 days)
  5-item scale, range 1 (strongly disagree) to (strongly agree). Weiner, B.J., Lewis, C.C., Stanick, C. et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Sci 12, 108 (2017). https://doi.org/10.1186/s13012-017-0635-3
Acceptability of the Intervention Scale | At the end of each cycle (each cycle is 42 days)
  5-item scale, range 1 (strongly disagree) to (strongly agree). Weiner, B.J., Lewis, C.C., Stanick, C. et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Sci 12, 108 (2017). https://doi.org/10.1186/s13012-017-0635-3
Appropriateness of the Intervention Scale | At the end of each cycle (each cycle is 42 days)
  5-item scale, range 1 (strongly disagree) to (strongly agree). Weiner, B.J., Lewis, C.C., Stanick, C. et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Sci 12, 108 (2017). https://doi.org/10.1186/s13012-017-0635-3

SECONDARY OUTCOMES:
Recruitment | At the end of each cycle (each cycle is 42 days)
  12-15 participants enrolled
Intervention Fidelity- participant characteristics | At the end of each cycle (each cycle is 42 days)
  proportion of participants are potentially PrEP eligible Black women (benchmark: 100%)
Intervention Fidelity | At the end of each cycle (each cycle is 42 days)
  Proportion of assigned materials distributed and assigned activities implemented (benchmark: 100%)
Acceptability of the intervention delivery | At the end of each session
  10-point scale assessment of facilitator performance. Benchmark: average acceptability rating of >7.5/10
Participant Enrollment | At the end of each cycle (each cycle is 42 days)
  Number of in-person participants in attendance at the first session. Benchmark: N = 12 - 15 in attendance at first session
Participant Retention | At the end of each cycle (each cycle is 42 days)
  Proportion of Session 1 participants who complete session 6. Benchmark: 80%
Feasibility of delivering 6 sessions in 6 weeks | At the end of each cycle (each cycle is 42 days)
  Delivery of intervention sessions according to the planned timeline (6 weeks)
Visual confirmation of self-reported PrEP uptake | At the end of each cycle (each cycle is 42 days)
  Photo confirmation of self-reported PrEP use.
Post-Intervention Follow-up | At the end of each cycle (each cycle is 42 days)
  Proportion of post-intervention surveys completed. Benchmark: 80%

CONTACTS AND LOCATIONS:
Overall Officials: Shawnika Hull, PhD, Principal Investigator — Rutgers University School of Communication and Information
Locations (2):
- United States (2):
  - The Women's Collective, Washington D.C., District of Columbia
  - Rutgers University, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No
As of now, there are no plans to share the IPD.